CLINICAL TRIAL: NCT02333409
Title: Electroacupuncture Analgesia in Patients With Inoperable Pancreatic Cancer: A Randomized, Sham-controlled Study
Brief Title: Acupuncture for Pain Control in Patients With Inoperable Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expertise resigned
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EA_CA pancreas
Record Dates: First submitted 2014-12-23; First posted 2015-01-07 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Cancer of Pancreas; Pain
Keywords: Cancer of pancreas; Acupuncture; Pain
MeSH Terms: conditions — Pancreatic Neoplasms; Pain | interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Active Comparator): A Hong Kong registered Chinese Medicine practitioner will give Electroacupuncture treatments. Patients will be treated in a comfortable prone position. Jiaji (Ex-B2) points form T8 to T12 bilaterally are chosen based on traditional Chinese medicine (TCM) theory and neurophysiologic basis of Jiaji points. After De Qi sensation is achieved, the handles of needles on homolateral T8-T12 Jiaji are respectively connected to the Han's acupoint nerve stimulator at a frequency of 2/100 Hz and a current of 1 mA with a disperse-dense waveform. The needles remained for 30 min. The treatment was given twice weekly on week 1 and week 3.
  Interventions: Procedure: Electroacupuncture
- Sham (Sham Comparator): For placebo acupuncture, sham placebo acupuncture needles (DongBang AcuPrime Acupuncture Inc., South Korea) will be used. Its validity and credibility have been well demonstrated. The needles with blunt tips are quickly put onto the same points used in the electroacupuncture group without inserting into the skin. The needles on homolateral T8 and T12 Jiaji are then connected to the electric stimulator, but with zero frequency and electric current.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Electroacupuncture (EA) has been used as a part of Traditional Chinese Medicine (TCM) and the benefits and success of EA as a viable treatment option for acute and chronic pain of various origins have been well-recognised.electro-acupuncture (EA) is taken place as to give out the stimulation with fixed frequency, pulse width and current to acupuncture needle for further promotion of analgesics effects.
  Other Names: Acupuncture

SUMMARY:
Pancreatic cancer is the sixth most common cause of cancer death in Hong Kong. Patients suffering from pancreatic cancer are associated with a poor prognosis and survival of less than one year is expected in inoperable tumours (1). Management of these patients would be towards palliation of symptoms. Severe pain occurs in 50 to 70% of the patients and this "intractable" pain is often difficult to treat (2). Pain management is a major part of the comprehensive therapy in patients with pancreatic cancer, and it also affects their quality of life. Electroacupuncture seems to be a promising way to control the cancer pain and reduce the dose and side effects of pain killers including opioid. This study aimed to investigate the efficacy and safety of electroacupuncture in reducing pancreatic cancer pain in patients suffering from inoperable pancreatic cancer.

DETAILED DESCRIPTION:
Patients suffering from pancreatic cancer are associated with a poor prognosis and survival of less than one year is expected in inoperable tumours. Management of these patients would be towards palliation of symptoms. Severe pain occurs in 50 to 70% of the patients and this "intractable" pain is often difficult to treat. Pain management is a major part of the comprehensive therapy in patients with pancreatic cancer, and it also affects their quality of life. Different pharmacological agents have been used in the past to control this pain and these include non-steroidal anti-inflammatory drugs and narcotic agents. However, these agents are associated with their own adverse effects and may further impair quality of life. Radiotherapy and celiac plexus neurolysis also can relieve the cancer pain, patients' responses are often variable and difficult to predict.

Recently, more and more studies were focused on the acupuncture for cancer pain. Electroacupuncture (EA) analgesia seems to be a promising way to control the cancer pain and reduce the dose and side effects of analgesics. The latest review in 2012 showed that acupuncture might be an effective analgesic adjunctive method for cancer pain after concluding the results of 15 randomized-control trials. Nevertheless, studies focused on patients with pancreatic cancer and results from randomized trials are lacking.

This study aims to investigate the efficacy and effectiveness of EA analgesia for patients with inoperable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All patients ≥ 18 years old with cytology or histology confirmed pancreatic cancer
2. Abdominal pain typical for pancreatic cancer
3. Inoperability of pancreatic cancer as demonstrated by computed tomography (CT), positron emission tomography (PET) scan or endoscopic ultrasonography (EUS).
4. Informed consent available

Exclusion Criteria:

1. Patients who are allergic to the acupuncture needles
2. Coagulopathy (prolongation of prothrombin time > 18 sec, thrombocytopenia <80,000 platelets/ml)
3. Another cause for abdominal pain such as pseudocyst, ulcer or other intra-abdominal disorder
4. Had been treated by acupuncture for pancreatic cancer within 1 year
5. Potential patient noncompliance (refusing to follow schedule of events)
6. Active alcohol or other drug use or significant psychiatric illness
7. Expected survival less than 3 months
8. Unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
pain scores in numeric rating scale (NRS) | 1 Month after Procedure
  Pain Score

SECONDARY OUTCOMES:
Procedural discomfort | Day 0 after procedure
  Discomfort feeling on visual analog scale (from 0 which implies no discomfort at all, to 100 which implies the worst discomfort imaginable)
Willingness to repeat procedure | 1 Month after Procedure
  Patient's willingness to repeat the procedure
Morbidities related to the procedures | 1 Month after Procedure
  Morbidities related to the procedures
Quality of Life scores | 1 Month after Procedure
  Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery; The Chinese University of Hong Kong, Hong Kong, Hong Kong